CLINICAL TRIAL: NCT01375608
Title: An Extended Phase 2 Study of Decitabine in Subjects With High Risk Sickle Cell Disease
Brief Title: Decitabine for High-Risk Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110184; 11-H-0184
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Neutropenia; Sickle Cell Disease
Keywords: Neutropenia; Hemaglobin; Coagulation Disorders; Thrombocytosis; Red Blood Cells; Sickle Cell Disease
MeSH Terms: conditions — Neutropenia; Anemia, Sickle Cell; Hemostatic Disorders; Thrombocytosis | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- decitabine (Other): active treatment
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 0.2mg/kg (range, 0.05-0.3 mg/kg) 1-2X/wk for a period of 48 weeks. Dose and frequency will be determined by hematologic toxicity and the achievement of an HbF level of greater the or equal to 20 percent.

SUMMARY:
Background:

* In sickle cell disease (SCD), the proteins in the red blood cells that carry oxygen do not behave normally. In parts of the body where there are low levels of oxygen or where oxygen is used more, the sickle hemoglobin proteins may change shape and stick together. This causes the red cells to clump, which reduces blood flow. This leads to even lower oxygen levels and causes damage and/or pain.
* One way to stop the red blood cells from sticking together is to increase the levels of fetal (baby or good ) hemoglobin. The good hemoglobin then takes the place of the sickle hemoglobin.
* Hydroxyurea is the only approved drug for SCD. But hydroxyurea works in only about two-thirds of people with SCD. Even in those cases it sometimes stops working over time.
* Researchers are interested in testing decitabine. The drug may help to increase fetal hemoglobin levels. But it has not yet been approved to treat SCD.

Objectives:

- To test the safety and effectiveness of decitabine in increasing fetal hemoglobin levels and improving the symptoms of sickle cell disease.

Eligibility:

- People at least 18 years of age who have sickle cell disease that has not improved after at least 6 months of hydroxyurea therapy. Those who cannot take hydroxyurea because of side effects may also participate.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests, a lung function test, and other tests as required.
* Participants will receive decitabine injections up to twice a week for 1 year. Depending on the response to treatments, the dose will remain the same or be reduced to once a week.
* Participants will be monitored with frequent blood tests and other studies as directed by the study doctors.
* After the study is completed, participants will go back to their usual sickle cell care. If decitabine has improved a participant's SCD, treatment may be continued under regular health coverage insurance if this can be arranged.

DETAILED DESCRIPTION:
Overview: Elevated fetal hemoglobin (HbF), whether pharmacologically induced or congenital, has a favorable impact on the morbidity and mortality of SCD. The agent currently used to elevate HbF, hydroxyurea (HU), has limited efficacy. There are mechanistic reasons to believe that the DNA methyltransferase inhibitor 5-aza-2 -deoxycytidine (decitabine) can more potently increase HbF. This has been demonstrated in vivo in animals and small phase 1/2 studies of decitabine in SCD subjects. Decitabine at low, non-cytotoxic doses was very well tolerated and very efficacious at increasing HbF and total hemoglobin (Hb) in subjects who did not respond to, or were intolerant of, HU. In addition to HbF levels, major improvements were noted in a range of surrogate clinical endpoints measuring red blood cell (RBC) adhesion, endothelial damage, and coagulation pathway activity. Also, substantial clinical improvement was seen in severely ill patients treated off-label. The primary objective herein is to provide evidence and guidance for a phase III study by demonstrating the dose and schedule of decitabine that when given over a 12 month period, produces sustained elevations in HbF without significant toxicity. Secondary objectives examine patient reported outcome measurements (PROMIS), crisis frequency, and laboratory indices that measure different domains of sickle cell pathophysiology and DNA methylation. These secondary and scientific measurements will be correlated with each other and examined over time to understand mechanisms of disease and the mechanism of action of the study drug.

Intervention: Decitabine starting dose of 0.2 mg/kg (range, 0.05-0.3 mg/kg) 1-2x/wk x 48 weeks

Hypotheses:

In SCD subjects at risk of early death, non-cytotoxic DNMT1 depletion using a metronomic (frequent but intermittent) regimen of the nucleoside analogue decitabine directly antagonizes a mechanism of gamma-globin repression, and produces sustained, clinically significant HbF elevations.

Primary Objective: To measure, in high-risk SCD subjects, the effect of chronic metronomic subcutaneous (SQ) decitabine administration on HbF levels. These aims are achieved through the conduct of an extended, open-label, phase 2 study in subjects who remain at high risk of early mortality and morbidity despite HU therapy.

Secondary Objectives: To measure, in high-risk SCD subjects, the effect of chronic metronomic SQ decitabine administration on clinical and laboratory indices of safety, patient reported outcome measures (PROMIS), frequency of crises, SCD pathophysiologic activity (hemolysis, coagulation, platelet activation and inflammation), and molecular effects of study drug.

Criteria for Evaluation:

Primary Endpoint: the percentage change in HbF level from baseline to the average percent over the final 3 months of the study period (48 weeks).

Secondary Endpoints: clinical and laboratory assessment of safety, patient reported outcomes (PROMIS), frequency of crises, quantity of F cells and F cell subsets, measurements of hemolysis, coagulation, platelet activation, inflammation, endothelial damage, pulmonary arterial pressure, DNMT levels, global and beta-globin locus specific DNA methylation.

Study Design: This is an extended, single arm, open-label, phase II clinical trial.

Study Population: Adults with symptomatic SCD who are at high risk of early mortality despite greater than or equal to 6 months of HU therapy. Specifically, they still have: HbF <5 percent, OR 3 or more pain episodes per year requiring parenteral narcotics, OR 1 or more acute chest syndrome episodes, OR hemoglobin <9 g/dL and absolute reticulocyte count (ARC) less than or equal to 250,000/mm(3). Subjects who meet the above criteria for high risk but are unwilling or unable to tolerate HU are also eligible.

Clinical and Laboratory Evaluations:

Pre-treatment and every 2 weeks: CBC, chem 20 including LDH, and retic count

Pre-treatment and every 4 weeks: interim medical history & physical exam, HbF%, and pregnancy test

Pre-treatment and every 12 weeks: urinanalysis, percent F-cells & percent F-reticulocytes, biomarkers, scientific correlative studies of DNA methylation

Pre-treatment, 24 and 48 weeks: PROMIS, PFT, 6 minute walk, endo-PAT

Pre-treatment and 48 weeks: erythropoietin level

Follow-ups every 3-4 months between 52-54 weeks and 93-96 weeks: interim medical history & physical exam, CBC, reticulocyte count, HbF percent, chem 20 (including LDH), and pregnancy test

Sample Size: 40 subjects

Data Analyses: The effect of decitabine on HbF levels over time will be explored using a general linear mixed model from which the average percent change from baseline to the average HbF level on the final 3 months of treatment will be estimated along with a 95 percent confidence interval. AE and other safety measurements will be summarized by age group, dose, and dose frequency at the time of AE onset. No interim analyses will be performed in this study.

Human Subjects: There is a risk of neutropenia, thrombocytosis, and teratogenicity. Patients must take precautions to use contraception and avoid pregnancy during treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects who meet all of the following criteria are eligible for enrollment into the study:

1. Age 18 years or older.
2. Written, informed consent provided by the subject before study entry.
3. Confirmed SCD (SS, S-beta (0)-thalassemia, or SC on hemoglobin electrophoresis),
4. Symptomatic SCD while on 6 months of HU OR symptomatic SCD and intolerant of HU (unable or unwilling to tolerate HU due to hematological or other toxicities). Symptomatic SCD is defined as having one of following:

   * HbF <5 percent, OR
   * 3 or more pain episodes per year requiring parenteral narcotics, OR
   * 1 or more acute chest syndrome episodes, OR
   * Hemoglobin <9 degree g/dL and ARC less than or equal to 250,000/mm(3),
5. Subject is in his/her steady state and not amidst any acute complication due to SCD.
6. Willing to use 2 forms of contraception. Some acceptable combinations include male partner using condoms and female partner using oral contraceptives, male partner using condoms and female partner who had bilateral oophorectomy, male partner who had a vasectomy and female partner using injectable contraceptives (e.g. Depo Provera).

EXCLUSION CRITERIA:

Since the protocol targets an at risk population, and the tolerability and potential benefits of this approach have been suggested in off-label treatment of seriously ill SCD patients, the exclusion criteria are not overly stringent and are primarily directed at avoiding teratogenic risks.

Subjects who meet any of the following criteria are disqualified from enrollment in the study:

1. Inability to give informed consent.
2. Experienced severe sepsis or septic shock within the previous 12 weeks.
3. Last HU or erythropoietin dose obtained within the previous 4 weeks. Renal replacement doses of erythropoietin is allowed as decitabine would not be expected to exert a red cell and/or HbF response when there is no endogenous erythropoietin production.
4. Participant is on chronic transfusion therapy (e.g., for history of TIA or stroke) and medically contraindicated to discontinue transfusions.
5. Currently pregnant or breast-feeding.
6. Sexually active female of childbearing potential (all females except those who are menopausal [appropriate age and no period for more than 12 months] or have had a hysterectomy and/or bilateral oophorectomy) who is unwilling to use at least 2 acceptable methods of contraception as determined by the investigators. The use of a condom by a male partner would be considered one acceptable method of contraception.
7. Sexually active male whose partner is of child-bearing potential and who is unwilling to use at least 2 acceptable methods of contraception as determined by the investigators during treatment and for 8 weeks after the last dose of decitabine.
8. Moribund or any concurrent disease (e.g., hepatic, renal, cardiac, metabolic) of such severity that death within 24 weeks is likely.
9. Other experimental or investigational drug therapy in the past 28 days.
10. Inability to bring ANC above 2 x 10(9) cells/L or platelet count less than 1,000 x 10(9) cells/L.

For female participants: Not having heterosexual sexual contact starting 4 weeks before beginning to take decitabine and continuing until 4 weeks after the last dose of decitabine OR using TWO methods of birth control. One birth control method must be highly effective, such as an Intrauterine Device (IUD), birth control pills, Depo-Provera (medroxyprogesterone acetate) injections, or tying of the fallopian tubes. The other additional effective method of birth control can be use of a diaphragm or a condom by the male partner. Birth control should begin at the screening visit and continue until 4 weeks after the last dose of decitabine. These steps must be taken even if the patient has a history of infertility, unless the patient has had a hysterectomy or has not had periods for at least 24 months.

For male participants: during decitabine treatment and 8 weeks after last dose of drug, a condom must be used when engaging in any sexual contact with a woman of child-bearing age, even in patients who have had a successful vasectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Hsieh, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] WATSON J. The significance of the paucity of sickle cells in newborn Negro infants. Am J Med Sci. 1948 Apr;215(4):419-23. doi: 10.1097/00000441-194804000-00008. No abstract available. PMID 18107723
- [Background] CONLEY CL, WEATHERALL DJ, RICHARDSON SN, SHEPARD MK, CHARACHE S. Hereditary persistence of fetal hemoglobin: a study of 79 affected persons in 15 Negro families in Baltimore. Blood. 1963 Mar;21:261-81. No abstract available. PMID 14022587
- [Background] Perrine RP, Pembrey ME, John P, Perrine S, Shoup F. Natural history of sickle cell anemia in Saudi Arabs. A study of 270 subjects. Ann Intern Med. 1978 Jan;88(1):1-6. doi: 10.7326/0003-4819-88-1-1. PMID 619731
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-H-0184.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Subcutaneous Decitabine in Sickle Cell Disease: decitabine (starting dose of 0.20 mg/kg, 2 days per week) to induce fetal hemoglobin (HbF) in patients with sickle cell anemia who are refractory to or intolerant of hydroxyurea
Period: Overall Study
Arm/Group | Subcutaneous Decitabine in Sickle Cell Disease
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Subcutaneous Decitabine in Sickle Cell Disease
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
total hemoglobin [Mean (Full Range); unit: g/dL] | 8.14 [4.9 to 12]
fetal hemoglobin [Mean (Full Range); unit: %] | 4.8 [1 to 13.5]

OUTCOME MEASURES:

1. Primary Outcome: The Percentage Change in HbF Level From Baseline to the Average Over the Final 1 Month of Study.
Time Frame: Final 1 month of study
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Decitabine in Sickle Cell Disease
Number analyzed (Participants) | 8
Participants
  total Hgb increase by >1g/dL AND HbF by >10% | 1
  total hgb increase by >1 g/dL OR HbF by 10% | 1
  total hgb increase by <1 g/dL OR HbF by <10% | 6

ADVERSE EVENTS:
Time Frame: January 2012 to December 2015
Arm/Group | Subcutaneous Decitabine in Sickle Cell Disease
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Decitabine in Sickle Cell Disease (N=10)
Sickle related (Musculoskeletal and connective tissue disorders) | 7 (30)
non sickle related SAE (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Decitabine in Sickle Cell Disease (N=10)
related to subcutaneous injection (Skin and subcutaneous tissue disorders) | 10 (10)
temporary musckle weakness with injection (Musculoskeletal and connective tissue disorders) | 4 (6)
rash (Skin and subcutaneous tissue disorders) | 5 (9)
GI disturbances (Gastrointestinal disorders) | 5 (10) — Nausea, vomiting, diarrhea, changes in appetite
headache (Musculoskeletal and connective tissue disorders) | 5 (5)
palpitation (Cardiac disorders) | 2 (3)
ENT (Ear and labyrinth disorders) | 5 (10) — metallic taste, hearing changes, jaw pain, dry mouth

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No